CLINICAL TRIAL: NCT02223429
Title: Biological Bases of Individual Variation in Paternal Nurturance
Brief Title: Neurobiological Bases of Paternal Nurturance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: James K. Rilling, PhD (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, James K. Rilling, PhD, Associate Professor, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB00044782; R21HD078778 (NIH)
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: Paternal nurturance; Oxytocin; Vasopressin; fMRI; Neurobiology
MeSH Terms: conditions — Diabetes Insipidus | interventions — Oxytocin; Vasopressins; Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- OT + placebo (Experimental): The OT + placebo group will self-administer no more than 1 ml solution of oxytocin or placebo in each nostril; five (5) sprays per each nostril, for a total of ten (10) sprays. The order of administration of drug and placebo will counterbalanced across subjects, such that half will receive OT first, and half will receive OT second.
  Interventions: Drug: Oxytocin; Drug: Placebo
- AVP + placebo (Experimental): The AVP + placebo group will self-administer no more than 1 ml solution of vasopressin or placebo in each nostril; five (5) sprays per each nostril, for a total of ten (10) sprays. The order of administration of drug and placebo will counterbalanced across subjects, such that half will receive AVP first, and half will receive AVP second.
  Interventions: Drug: Vasopressin; Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 1 ml solution in each nostril; five (5) sprays per each nostril, for a total of ten (10) sprays
  Other Names: Pitocin; Syntocinon; OT
  Arms: OT + placebo
Drug: Vasopressin — 1 ml solution in each nostril; five (5) sprays per each nostril, for a total of ten (10) sprays
  Other Names: Argipressin; Arginine vasopressin (AVP); Antidiuretic hormone (ADH)
  Arms: AVP + placebo
Drug: Placebo — 1 ml solution in each nostril; five (5) sprays per each nostril, for a total of ten (10) sprays

SUMMARY:
The overall goal of this project is to identify the genetic, hormonal, and neurobiological influences on paternal nurturing behavior and to determine if fathers' neural responses to infants can be modulated by neuropeptides known to play a role in parenting in experimental animal models.

The aim is to determine if pharmacological manipulation of central oxytocin (OT) and vasopressin (AVP) levels influences the neural response to viewing pictures of one's own infant or to hearing cry stimuli. In a double-blind procedure, fathers with 1-3 year old children will be scanned on two separate occasions; once under the influence of OT/AVP and once under the influence of placebo. Fathers will be randomized to either OT or AVP, and order of administration of drug and placebo will counterbalanced across subjects. Fathers will be scanned while viewing pictures of their own and an unknown child and while listening to unknown infant cry stimuli.

The investigators hypothesize:

* OT will augment the ventral tegmental area (VTA), ventral striatum and medial orbitofrontal cortex (mOFC) response to viewing pictures of one's own child, and will augment the primary auditory cortex (AI) response of fathers to infant cries.
* AVP will augment the lateral septum response to viewing own child pictures.

DETAILED DESCRIPTION:
30 fathers of children aged 1-3 will participate in two functional imaging sequence (fMRI) sessions, once under the influence of OT/AVP, and once under the influence of placebo. Fathers will be restricted to men who are living with their biological child and an adult partner (male or female) that they are in a committed relationship with. All fathers will receive two fMRI scans on two different occasions, separated by 2-10 days. 15 fathers will be randomized to intranasal OT, the other 15 will be randomized to intranasal AVP. Within each drug group, the order of administration of drug and placebo will counterbalanced across subjects, such that 15 will receive OT/AVP first, and 15 will receive OT/AVP second. During the fMRI scans, fathers will view pictures of their own and unknown children, as well as unknown adults. Afterwards, while still in the scanner, they will listen to infant cry and control stimuli. After exiting the scanner, fathers will again listen to the cry stimuli and will rate their emotional reaction to the cry stimuli on the following dimensions using a 7 point likert scale: irritated, sympathetic, alarmed, angry, upset, compassionate, distressed, annoyed, and tender.

ELIGIBILITY:
Inclusion Criteria:

* above 18
* biological fathers of 1-3 year old infants who are currently cohabitating with the child's mother
* normal or corrected-to-normal vision of 20/40

Exclusion Criteria:

* current or past history of mental illness
* active medical or neurological disorder
* current or past history of alcohol or drug dependence
* claustrophobic (at the discretion of the PI with subject consultation)
* history of seizures or other neurological disorder
* history of hypertension, cardiovascular disease, nephritis, diabetes or other endocrine diseases or malignancy
* ferrous metal in any part of the body
* history of asthma or migraine headaches (can be included at the discretion of the study physician or nurse practitioner if episodes are infrequent and no active problems at time of study, not medicated)
* history of head trauma or psychiatric illness, as well as those who are receiving or have received over the past year, medication with known psychoactive effects (included at the discretion of the PI as these are exclusion criteria due to data quality concerns and not safety concerns; head trauma should be minimal enough deemed by the PI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James K Rilling, Ph.D., Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital, Atlanta, Georgia
  - Emory University 1462 Clifton Rd, Atlanta, Georgia

REFERENCES:
- [Background] Hamann S, Herman RA, Nolan CL, Wallen K. Men and women differ in amygdala response to visual sexual stimuli. Nat Neurosci. 2004 Apr;7(4):411-6. doi: 10.1038/nn1208. Epub 2004 Mar 7. PMID 15004563
- See also: Related Info — http://anthropology.emory.edu/home/people/faculty/rilling.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place from 9/29/2014 through 2/3/2016.
Pre-assignment Details: Of the 35 participants consented for participation, 32 began the study. Three participants were lost to follow up after signing the consent form.
Groups:
- OT First, Followed by Placebo: Participants were randomized to receive no more than 1 ml solution of self-administered oxytocin spray in each nostril followed by no more than 1 ml solution of self-administered placebo spray in each nostril. Time between interventions was 2-10 days.
- Placebo First, Followed by OT: Participants were randomized to receive no more than 1 ml solution of self-administered placebo spray in each nostril followed by no more than 1 ml solution of self-administered oxytocin spray in each nostril. Time between interventions was 2-10 days.
- AVP First, Followed by Placebo: Participants were randomized to receive no more than 1 ml solution of self-administered vasopressin spray in each nostril followed by no more than 1 ml solution of self-administered placebo spray in each nostril. Time between interventions was 2-10 days.
- Placebo First, Followed by AVP: Participants were randomized to receive no more than 1 ml solution of self-administered placebo spray in each nostril followed by no more than 1 ml solution of self-administered vasopressin spray in each nostril. Time between interventions was 2-10 days.
Period: Overall Study
Arm/Group | OT First, Followed by Placebo | Placebo First, Followed by OT | AVP First, Followed by Placebo | Placebo First, Followed by AVP
Started | 8 | 8 | 8 | 8
Completed | 7 | 8 | 8 | 8
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only participants who completed the study were included in the baseline analysis. Among the 32 subjects who started the study, one participant did not complete MRI scanning and was not included in any data analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | OT First, Followed by Placebo | Placebo First, Followed by OT | AVP First, Followed by Placebo | Placebo First, Followed by AVP | Total
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.14 (4.14) | 31.88 (4.61) | 32.25 (5.75) | 34 (4.75) | 32.81 (4.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 7 | 8 | 8 | 8 | 31
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 8 | 8 | 31

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Signal Change in Ventral Tegmental Area (VTA)
Description: The effect of the drug will be assessed by determining changes in brain activation to own child pictures versus adult pictures (O-A) between OT treatment and placebo treatments (OT-PL) from functional magnetic resonance imaging (fMRI). Changes will be assessed in the OT group only per protocol.
Time Frame: Baseline, Visit 2 (Up to 10 days)
Population: The analysis was completed per protocol for the OT + placebo groups only.
Measure: Mean (Standard Deviation); unit: Percent signal change
Groups:
- Oxytocin: Participants were randomized to receive no more than 1 ml solution of self-administered oxytocin spray in each nostril followed by no more than 1 ml solution of self-administered placebo spray in each nostril. Time between interventions was 2-10 days.
- Placebo: Participants were randomized to receive no more than 1 ml solution of self-administered placebo spray in each nostril followed by no more than 1 ml solution of self-administered oxytocin spray in each nostril. Time between interventions was 2-10 days.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 15 | 15
Percent signal change | 0.54 (1.24) | 0.27 (1.34)

2. Primary Outcome: Mean Percent Signal Change in Right Ventral Striatum
Description: as for outcome 1
Time Frame: Baseline, Visit 2 (Up to 10 days)
Population: The analysis was completed per protocol for the OT + placebo groups only.
Measure: Mean (Standard Deviation); unit: Percent signal change
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 15 | 15
Percent signal change | -1.28 (1.59) | -0.81 (1.74)

3. Primary Outcome: Mean Percent Signal Change in Right Medial Orbitofrontal Cortex
Description: as for outcome 1
Time Frame: Baseline, Visit 2 (Up to 10 days)
Population: The analysis was completed per protocol for the OT + placebo groups only.
Measure: Mean (Standard Deviation); unit: Percent signal change
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 15 | 15
Percent signal change | -0.22 (0.64) | -0.53 (0.96)

4. Primary Outcome: Mean Percent Signal Change in Caudate Nucleus
Description: The effect of the drug will be assessed by determining changes in brain activation to own child pictures versus adult pictures (O-A) between OT treatment and placebo treatments (OT-PL) from functional magnetic resonance imaging (fMRI).
Time Frame: Baseline, Visit 2 (Up to 10 days)
Population: The analysis was completed per protocol for the OT + placebo groups only.
Measure: Mean (Standard Deviation); unit: Percent signal change
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 15 | 15
Percent signal change | 0.85 (0.92) | -0.27 (0.67)

5. Primary Outcome: Mean Percent Signal Change in the Visual Cortex
Description: as for outcome 4
Time Frame: Baseline, Visit 2 (Up to 10 days)
Population: The analysis was completed per protocol for the OT + placebo groups only.
Measure: Mean (Standard Deviation); unit: Percent signal change
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 15 | 15
Percent signal change | 0.83 (1.18) | 0.10 (1.34)

6. Primary Outcome: Mean Percent Signal Change in the Anterior Cingulate Cortex
Description: as for outcome 4
Time Frame: Baseline, Visit 2 (Up to 10 days)
Population: Analysis was conducted in the OT+placebo groups only.
Measure: Mean (Standard Deviation); unit: Percent signal change
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 15 | 15
Percent signal change | 0.27 (0.60) | -0.39 (0.63)

7. Secondary Outcome: Change in Plasma Levels of Vasopressin (AVP)
Description: Peripheral levels of AVP will be assessed via assay of plasma collected.
Time Frame: Baseline, Visit 2 (Up to 10 days)
Population: Zero participants were analyzed as AVP samples were not assayed.
Groups:
- AVP + Placebo: The AVP + placebo group self-administered no more than 1 ml solution of vasopressin or placebo in each nostril; five (5) sprays per each nostril, for a total of ten (10) sprays. The order of administration of drug and placebo was counterbalanced across subjects, such that half received AVP first, and half received AVP second.
Arm/Group | AVP + Placebo
Number analyzed (Participants) | 0

8. Secondary Outcome: Change in Plasma Levels of Oxytocin (OT)
Description: Peripheral levels of OT will be assessed via assay of plasma collected.
Time Frame: Baseline, Visit 2 (Up to 10 days)
Population: Zero participants were analyzed as samples were not assayed.
Groups:
- OT + Placebo Group: The OT + placebo group self-administered no more than 1 ml solution of oxytocin or placebo in each nostril; five (5) sprays per each nostril, for a total of ten (10) sprays. The order of administration of drug and placebo was counterbalanced across subjects, such that half received OT first, and half received OT second.
Arm/Group | OT + Placebo Group
Number analyzed (Participants) | 0

9. Secondary Outcome: Difference in Cry Rating Scores Between OT and Placebo
Description: The effect of the drug will be assessed by analyzing the differences between ratings of infant cries under OT and placebo treatment on a 7-point likert scale. Sixteen adjectives will be used to describe two different cries. Participants will rate each cry from 1-7 where one represents "not at all" and 7 represents "extremely". Difference is defined as OT minus placebo scores.
Time Frame: Baseline, Visit 2 (Up to 10 days)
Population: Of the 15 participants who were administered oxytocin in combination with placebo at any time point during the study, data were analyzed for 14 participants. One participant was excluded from the analysis due to missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Oxytocin: All participants who were administered oxytocin at any time point during the study and have completed the cry rating scale.
- Placebo: All participants who were administered placebo at any time point during the study and have completed the cry rating scale.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 14 | 14
units on a scale
  Cry 1 Grating | 3.71 (1.90) | 4.64 (1.60)
  Cry 1 Urgent | 4.29 (1.94) | 4.86 (1.66)
  Cry 1 Piercing | 4.29 (1.86) | 4.36 (1.78)
  Cry 1 Aversive | 3.57 (1.74) | 3.36 (1.45)
  Cry 1 Compelling | 4.57 (1.79) | 5.00 (1.92)
  Cry 1 Manipulative | 2.86 (1.92) | 2.29 (1.38)
  Cry 1 Spoiled | 2.14 (1.10) | 2.07 (.92)
  Cry 1 Irritated | 3.07 (1.86) | 3.29 (1.98)
  Cry 1 Sympathetic | 4.71 (1.50) | 4.43 (1.65)
  Cry 1 Alarmed | 4.21 (2.00) | 4.07 (2.20)
  Cry 1 Angry | 2.43 (1.83) | 2.57 (1.79)
  Cry 1 Upset | 3.07 (1.90) | 3.29 (2.30)
  Cry 1 Compassionate | 4.86 (2.07) | 5.14 (1.56)
  Cry 1 Distressed | 3.57 (2.24) | 3.64 (1.91)
  Cry 1 Annoyed | 2.43 (1.65) | 2.43 (1.51)
  Cry 1 Tender | 3.79 (1.63) | 3.64 (1.82)
  Cry 2 Grating | 3.43 (2.17) | 3.79 (1.93)
  Cry 2 Urgent | 4.93 (1.54) | 4.43 (2.07)
  Cry 2 Piercing | 3.71 (2.23) | 4.00 (2.32)
  Cry 2 Aversive | 3.50 (1.83) | 4.07 (1.39)
  Cry 2 Compelling | 5.21 (1.37) | 5.14 (1.56)
  Cry 2 Manipulative | 2.43 (2.03) | 2.36 (1.74)
  Cry 2 Spoiled | 2.00 (1.41) | 2.00 (1.36)
  Cry 2 Irritated | 2.21 (1.53) | 2.36 (1.69)
  Cry 2 Sypmathetic | 5.86 (1.17) | 5.64 (1.45)
  Cry 2 Alarmed | 4.36 (2.34) | 4.57 (2.17)
  Cry 2 Angry | 1.79 (1.05) | 1.79 (.98)
  Cry 2 Upset | 2.86 (1.56) | 2.57 (1.40)
  Cry 2 Compassionate | 5.71 (1.49) | 5.43 (1.70)
  Cry 2 Distressed | 3.36 (2.17) | 3.86 (2.21)
  Cry 2 Annoyed | 2.00 (1.30) | 1.93 (1.44)
  Cry 2 Tender | 4.50 (1.22) | 4.79 (1.48)

10. Secondary Outcome: Difference in Cry Rating Scores Between AVP and Placebo
Description: The effect of the drug will be assessed by analyzing the differences between ratings of infant cries under AVP and placebo treatment on a 7-point likert scale. Sixteen adjectives will be used to describe two different cries. Participants will rate each cry from 1-7 where one represents "not at all" and 7 represents "extremely". Difference is defined as AVP minus placebo scores.
Time Frame: Baseline, Visit 2 (Up to 10 days)
Population: Analysis was completed according to protocol for all participants who were administered AVP in combination with placebo at any time point during the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Vasopressin (AVP): All participants who were administered AVP at any time point during the study and have completed the cry rating scale.
Arm/Group | Vasopressin (AVP) | Placebo
Number analyzed (Participants) | 16 | 16
units on a scale
  Cry 1 Grating | 4.69 (1.45) | 4.06 (1.611)
  Cry 1 Urgent | 5.44 (1.09) | 5.31 (1.01)
  Cry 1 Piercing | 4.81 (1.47) | 4.19 (1.33)
  Cry 1 Aversive | 3.94 (1.48) | 3.81 (1.38)
  Cry 1 Compelling | 4.56 (1.32) | 5.00 (1.21)
  Cry 1 Manipulative | 3.06 (1.48) | 2.69 (1.49)
  Cry 1 Spoiled | 2.44 (1.03) | 1.94 (1.06)
  Cry 1 Irritated | 3.44 (1.82) | 3.44 (1.86)
  Cry 1 Sympathetic | 5.06 (1.81) | 4.38 (2.09)
  Cry 1 Alarmed | 4.88 (1.46) | 4.38 (1.41)
  Cry 1 Angry | 1.94 (1.44) | 1.81 (1.22)
  Cry 1 Upset | 3.00 (1.55) | 2.63 (1.20)
  Cry 1 Compassionate | 4.88 (1.71) | 4.94 (1.65)
  Cry 1 Distressed | 3.31 (1.35) | 3.31 (1.58)
  Cry 1 Annoyed | 2.50 (1.67) | 2.25 (1.48)
  Cry 1 Tender | 4.00 (1.51) | 4.19 (1.56)
  Cry 2 Grating | 3.25 (1.69) | 3.38 (1.78)
  Cry 2 Urgent | 5.13 (1.26) | 5.25 (0.78)
  Cry 2 Piercing | 3.13 (1.10) | 3.56 (1.50)
  Cry 2 Aversive | 3.44 (1.55) | 3.44 (1.09)
  Cry 2 Compelling | 4.50 (1.63) | 5.00 (0.97)
  Cry 2 Manipulative | 2.63 (2.06) | 2.38 (1.46)
  Cry 2 Spoiled | 2.19 (1.33) | 2.31 (1.40)
  Cry 2 Irritated | 2.13 (1.50) | 2.63 (1.46)
  Cry 2 Sypmathetic | 4.88 (1.75) | 4.94 (1.69)
  Cry 2 Alarmed | 4.31 (1.74) | 4.25 (1.69)
  Cry 2 Angry | 2.13 (1.63) | 2.00 (1.16)
  Cry 2 Upset | 3.19 (1.91) | 2.88 (1.59)
  Cry 2 Compassionate | 4.88 (1.75) | 4.75 (1.84)
  Cry 2 Distressed | 3.06 (1.77) | 3.06 (1.53)
  Cry 2 Annoyed | 2.19 (1.68) | 1.88 (1.26)
  Cry 2 Tender | 4.44 (1.10) | 4.50 (1.71)

11. Secondary Outcome: Mean Percent Signal Change in Primary Auditory Cortex
Description: as for outcome 1
Time Frame: Baseline, Visit 2 (Up to 10 days)
Population: The analysis was completed per protocol for the OT + placebo group only.
Measure: Mean (Standard Deviation); unit: Percent signal change
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 15 | 15
Percent signal change | 0.10 (0.15) | 0.10 (0.24)

12. Secondary Outcome: Mean Percent Signal Change in Right Lateral Septum
Description: The effect of the drug will be assessed by determining changes in brain activation to own child pictures versus adult pictures (O-A) between AVP treatment and placebo treatments (AVP-PL) from functional magnetic resonance imaging (fMRI). Changes will be assessed in the AVP group only per protocol.
Time Frame: Baseline, Visit 2 (Up to 10 days)
Population: The analysis was conducted in the AVP groups only per protocol. One person from each order of administration were excluded from the analysis due to motion issues in their imaging data.
Measure: Mean (Standard Deviation); unit: Percent signal change
Groups:
- Vasopressin (AVP): Participants were randomized to receive no more than 1 ml solution of self-administered vasopressin spray in each nostril followed by no more than 1 ml solution of self-administered placebo spray in each nostril. Time between interventions was 2-10 days.
- Placebo: Participants were randomized to receive no more than 1 ml solution of self-administered placebo spray in each nostril followed by no more than 1 ml solution of self-administered vasopressin spray in each nostril. Time between interventions was 2-10 days.
Arm/Group | Vasopressin (AVP) | Placebo
Number analyzed (Participants) | 14 | 14
Percent signal change | 0.19 (0.43) | 0.36 (0.56)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the study (2 years).
Groups:
- OT Treatment: The OT group self-administered no more than 1 ml solution of oxytocin in each nostril; five (5) sprays per each nostril, for a total of ten (10) sprays.
  This group also went through the Placebo of OT treatment.
- AVP Treatment: The AVP group self-administered no more than 1 ml solution of vasopressin in each nostril; five (5) sprays per each nostril, for a total of ten (10) sprays.
  This group also went through the Placebo of AVP treatment.
- Placebo of OT: The placebo of OT group self-administered no more than 1 ml solution of placebo of OT in each nostril; five (5) sprays per each nostril, for a total of ten (10) sprays.
  This group also went through the OT treatment.
- Placebo of AVP: The placebo of AVP group self-administered no more than 1 ml solution of placebo of AVP in each nostril; five (5) sprays per each nostril, for a total of ten (10) sprays.
  This group also went through the AVP treatment.
Arm/Group | OT Treatment | AVP Treatment | Placebo of OT | Placebo of AVP
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 3/16 | 2/16 | 0/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OT Treatment (N=16) | AVP Treatment (N=16) | Placebo of OT (N=16) | Placebo of AVP (N=16)
Claustrophobia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
High Blood Pressure prior to Drug Administration (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Headache prior to Drug Administration (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Spray Strength Intolerance (Product Issues) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Participants reported that the vasopressin nasal spray was too strong. The brand was subsequently changed.

LIMITATIONS AND CAVEATS:
Plasma levels of vasopressin (AVP) and peripheral levels of oxytocin (OT) were not assayed due to lack of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes